CLINICAL TRIAL: NCT03891030
Title: Effectiveness of Checklist Based Box System Interventions (CBBSI) on Improving Utilization of Maternal Health Service in North West, Ethiopia: a Cluster Randomized Controlled Trial
Brief Title: Checklist Based Box System Interventions
Acronym: CBBSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jimma University (Other)
Collaborators: Armauer Hansen Research Institute (AHRI) (Unknown)
Responsible Party: Principal Investigator, Netsanet Belete, Msc, Jimma University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CBBSI/2019
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Maternal Health Service

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Checklist Based Box system (Experimental): Pregnant mothers will receive scheduled person-centered health educations starting from: they are identified as suspected pregnant mother up to attending their third PNC visit. In between the first ANC and the third PNC drop out tracing mechanisms will be applied, for mothers who fail to utilize the recommended maternal health services.
  Interventions: Other: Checklist Based Box system intervention
- Routine maternal health care (No Intervention): Pregnant mothers in this arm will receive the usual routine maternal health care.

INTERVENTIONS:
Other: Checklist Based Box system intervention — The intervention has both behavioural change and service utilization drop out tracing mechanism. Special type of boxes designed to schedule health educations and continued service utilization monitoring boxes will be placed at health posts and health centers respectively. Community level survey will be conducted to identify suspected pregnant mothers using stanback et al, 1999 checklist, and mothers are linked to health centers. Then, they will be followed for their subsequent attendance of consecutive maternal health services (ANC 2nd-third PNC). Mothers who fail to utilize the service will be traced; will get person-centered health education to continue the service.
  Arms: Checklist Based Box system

SUMMARY:
Maternal mortality is still high in Ethiopia. Antenatal care (ANC), use of skilled delivery attendants and postnatal care (PNC) services are key maternal health care services that can significantly reduce maternal mortality. However, interventions applied to the continued utilization of these key maternal heath services in a continuum of care approach (i.e. early initiation of ANC and continued utilization up to four plus vists, health facility delivery attended by skilled health care providers and attending three PNC visits) were not well applied and studied.

Hence, the purpose of this study is to test the effectiveness of checklist based box system interventions on improving utilization of maternal health service (Antenatal care, skilled birth attendance and postnatal care) utilization.

DETAILED DESCRIPTION:
Cluster Randomized controlled trial study design will be employed. The sample size for this study was calculated based on the recommendations for sample size calculations for cluster randomized controlled trials with fixed number of clusters, by using STATA. The following assumptions were considered: to detect an increase of postnatal care three utilization from 16% to 28% from previous study, number of clusters available-30, with 95% confidence interval and 80% power, intra-cluster correlation coefficient of 0.04849 from similar studies, 15 clusters per arm. The sample size was calculated to determine number of observations required per cluster, for two-sample comparison of proportions (using normal approximation), Assuming individual randomization, sample size per arm is 194. Then allowing for cluster randomization, average cluster size required is 40, and the final sample size is 1200 pregnant mothers (600 in intervention, and 600 in control). Data analysis will take place in two levels (cluster and individual). Risk ration will be computed at cluster level, and the results of this cluster summary will be compared using t-test. Primary and secondary outcomes will be compared between intervention and control groups with random effects logistic regression models, taking account of clustering.

ELIGIBILITY:
Inclusion Criteria:

* Mothers residing in three of the selected districts Debre-Markos, Gozamin and Machakel districts Mother who are positive for Stanback et al, 1999 pregnancy screening criteria and found HCG positive (confirmed pregnancy) Gestational age of less than 16 weeks Mothers willing to participate in the study

Exclusion Criteria:

* Women who have severe psychological illness, which could interfere with, consent and study participation, Those who have sever clinical complications that need hospitalization Mothers who need special type of ANC follow-up, other than the recommended focused ANC

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Continued maternal health service utilization (ANC 1-4), Institutional Delivery, PNC (1-3) | 42 days after delivery
  Proportion of mothers receiving continued maternal health service (four ANC, skilled birth attendance and PNC three) in the intervention and control clusters, assessed using standard questionnaire

SECONDARY OUTCOMES:
Early Initiation of Antenatal care (Before 16 Weeks of Gestation) | 16 weeks of gestation
  Proportion of mothers attending ANC before 16 weeks of gestation in the intervention and control clusters, assessed using 4-visit WHO ANC Model
Attending four antenatal care follow up, (36-40 weeks of gestation) | 40 weeks of gestation
  Proportion of mothers attending the fourth ANC in the intervention and control clusters, assessed using 4-visit WHO ANC Model
Institutional delivery attended by skilled Birth attendance | after 40 weeks of gestation
  Proportion of mothers attending institutional delivery in the intervention and control clusters, assessed using standard questionnaire
Postnatal care follow-up (First 6 hours, 6 days and 6 weeks of delivery) | 42 days after delivery
  Proportion of mothers attending the third PNC in the intervention and control clusters: assessed using standard questionnaire
Knowledge towards maternal health service | 42 days after delivery
  Knowledge of mothers towards healthy pregnancy, delivery and the postnatal care period in the intervention and control clusters: assessed using Knowledge questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Netsanet Belete, Msc, Principal Investigator — Jimma University; Mulusew Gerbaba, PhD, Study Director — Jimma University; Gurmesa Tura, PhD, Study Director — Jimma University
Locations (1):
- East Gojjam zone, Debre Markos, Northwest, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Participant flow, outcome measure statistical analysis

REFERENCES:
- [Derived] Andargie NB, Debelew GT. Effectiveness of checklist-based box system intervention (CBBSI) versus routine care on improving utilization of antenatal care visits in Northwest Ethiopia: a cluster randomized controlled trial. BMC Health Serv Res. 2022 Apr 9;22(1):466. doi: 10.1186/s12913-022-07894-7. PMID 35397607
- [Derived] Andargie NB, Debelew GT. Effect of checklist based box system interventions on improving institutional delivery among reproductive age women in Northwest Ethiopia: generalized structural equation modeling. Arch Public Health. 2022 Jan 4;80(1):5. doi: 10.1186/s13690-021-00774-2. PMID 34983665
- [Derived] Andargie NB, Debelew GT. Effectiveness of checklist-based box system intervention (CBBSI) versus routine care on improving postnatal care utilization in Northwest Ethiopia: a cluster randomized controlled trial. Reprod Health. 2021 Nov 20;18(1):234. doi: 10.1186/s12978-021-01283-9. PMID 34801045
- [Derived] Andargie NB, Jebena MG, Debelew GT. Effectiveness of Checklist-Based Box System Interventions (CBBSI) versus routine care on improving utilization of maternal health services in Northwest Ethiopia: study protocol for a cluster randomized controlled trial. Trials. 2020 Feb 7;21(1):151. doi: 10.1186/s13063-019-4002-3. PMID 32033576